CLINICAL TRIAL: NCT00715793
Title: Phase I/II Trial of the Combination of Decitabine and Temozolomide in the Treatment of Patients With Metastatic Melanoma
Brief Title: Combination of Decitabine and Temozolomide in the Treatment of Patients With Metastatic Melanoma
Acronym: UPCI-07-008
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hussein Tawbi (Other)
Collaborators: Eisai Inc. (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, Hussein Tawbi, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 07-008
Record Dates: First submitted 2008-06-27; First posted 2008-07-15 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Malignant Melanoma
Keywords: Decitabine; Temozolomide; Metastatic; Melanoma; Non-resectable; Stage IIIB melanoma; stage IV melanoma; TMZ; DTIC; promoter methylation; skin cancer; chemotherapy
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Skin Neoplasms | interventions — Decitabine; Dacarbazine; Temozolomide; Biopsy; Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Decitabine; Drug: Temozolomide; Procedure: biopsy

INTERVENTIONS:
Drug: Decitabine — In Part I patients will be treated on a standard "3+3" phase I dose-escalation design starting at 0.075 mg/kg until a decitabine dose level of 0.15 mg/kg is reached, or, in case unacceptable toxicities are observed, at the maximum tolerated dose (Phase II recommended dose). Decitabine will be administered at the specified dose level, intravenously, daily 5 days a week for the first 2 weeks of a 6-week cycle.
  Other Names: DTIC
Drug: Temozolomide — Temozolomide is available in 25 mg and 100 mg tablets that will be administered orally; doses will be rounded to the nearest 25 mg. Temozolomide will be administered orally at 75 mg/m2 daily for 4 weeks starting on week 2 of a 6-week cycle.
  Other Names: TMZ
Procedure: biopsy — Fine needle aspirates (FNA) and/or core biopsies of tumor samples will be obtained from consenting patients with accessible, evaluable disease, on days 1, 8, 15, and 29 of the first cycle and when patients go off study. Biopsies are optional in Phase I and required for all consenting subjects in Phase II.
  Other Names: fine needle aspirate; FNA; core biopsy

SUMMARY:
The combination of TMZ and DAC may effect dual modulation of DNA repair genes resulting in improved clinical response.

DETAILED DESCRIPTION:
Primary Objectives:

* Phase I: To determine the safety, tolerability, and Phase II recommended dose of the combination of extended schedule TMZ and DAC.
* Phase II: To determine the efficacy, as measured by overall response rate, of the combination of extended schedule TMZ and DAC given at the Phase II recommended dose to patients with metastatic melanoma.

Secondary Objectives:

* To determine pharmacokinetics of the combination of TMZ and DAC in patients with metastatic melanoma.
* To determine, in peripheral blood mononuclear cells (PBMC) and tumor tissue, the pharmacodynamic effects of the combination of TMZ and DAC on promoter methylation and expression of selected genes and correlate these with response.
* To determine the progression-free survival of patients treated with the combination of TMZ and DAC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have non-resectable Stage IIIB or stage IV metastatic melanoma that have progressed despite prior therapies.
* Life expectancy of at least 12 weeks.
* ECOG performance status of 0, 1 and 2.
* ≥18 years of age.
* Patients who have not received any other chemotherapeutic, biological or investigational agent within 28 days of study drug administration.
* First line and active brain metastases (metastatic lesions to the brain that have been adequately treated with surgery and/or appropriate radiation therapy and that have documented stability for >4 weeks or >2 weeks if treated with stereotactic radiosurgery, remain eligible)

Exclusion Criteria:

* Any evidence of renal dysfunction (proteinuria, estimated creatinine clearance from serum creatinine test of <60 ml/min).
* Impaired hepatic function (liver enzymes greater than twice the upper limit of normal or bilirubin > 2.0 except in patients with Gilbert's syndrome).
* Prior treatment with alkylating agents (including TMZ and DTIC).
* Active brain metastases (metastatic lesions to the brain that have been adequately treated with surgery and/or appropriate radiation therapy and that have documented stability for >4 weeks remain eligible).
* Active infections or serious general medical conditions.
* Female patients of child-bearing age who are not on adequate contraception, or are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DAC (Decitabine) 0.075 mg/kg + TMZ (Temozolomide): Patients with non-resectable stage IIIB/C or stage IV metastatic melanoma with either no prior therapy or have progressed despite prior therapies, who were treated with DAC 0.075 mg/kg intravenously daily × 5 days/week for 2 weeks, TMZ orally 75 mg/m^2 qd for weeks 2-5 of a 6-week cycle.
- DAC (Decitabine) 0.15 mg/kg + TMZ (Temozolomide): Patients with non-resectable stage IIIB/C or stage IV metastatic melanoma with either no prior therapy or have progressed despite prior therapies, who were treated with DAC 0.15 mg/kg intravenously daily × 5 days/week for 2 weeks, TMZ orally 75 mg/m^2 qd for weeks 2-5 of a 6-week cycle.
Period: Phase 1 RP2D DAC + TMZ
Arm/Group | DAC (Decitabine) 0.075 mg/kg + TMZ (Temozolomide) | DAC (Decitabine) 0.15 mg/kg + TMZ (Temozolomide)
Started | 4 | 6
Completed | 3 | 6
Not Completed | 1 | 0
Not completed — secondary disease in Cycle 1 | 1 | 0
Period: Phase 2 DAC (0.15 mg/kg) + TMZ
Arm/Group | DAC (Decitabine) 0.075 mg/kg + TMZ (Temozolomide) | DAC (Decitabine) 0.15 mg/kg + TMZ (Temozolomide)
Started | 0 | 29
Completed | 0 | 27
Not Completed | 0 | 2
Not completed — not assessable for tumor response | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants DAC (Decitabine) + TMZ (Temozolomide): Patients with non-resectable stage IIIB/C or stage IV metastatic melanoma with either no prior therapy, or, have progressed despite prior therapies, who were treated with DAC 0.15 mg/kg intravenously daily × 5 days/week for 2 weeks + TMZ orally 75 mg/m^2 qd for weeks 2-5 of a 6-week cycle).
Arm/Group | All Study Participants DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 63.3 [36.2 to 77.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Experienced a Dose Limiting Toxicity (DLT)
Description: Dose-limiting toxicities (DLTs) were defined as grade 4 neutropenia or thrombocytopenia which lasts >7 days; grade 3 or 4 febrile neutropenia; grade 3 or greater non-hematological toxic effects.
Time Frame: Up to 26 months
Population: Patients participating in the Phase 1 portion of the study that were treated on a standard "3+3" phase I dose-escalation design who were observed for unacceptable toxicities.
Measure: Number; unit: percentage of participants
Groups:
- Dose Level 1:DAC (Decitabine) 0.075 mg/kg + TMZ (Temozolomide): Patients with non-resectable stage IIIB/C or stage IV metastatic melanoma with either no prior therapy or have progressed despite prior therapies, who were treated with DAC 0.075 mg/kg intravenously daily × 5 days/week for 2 weeks, TMZ orally 75 mg/m^2 qd for weeks 2-5 of a 6-week cycle.
- Dose Level 2:DAC (Decitabine) 0.15 mg/kg + TMZ (Temozolomide): Patients with non-resectable stage IIIB/C or stage IV metastatic melanoma with either no prior therapy or have progressed despite prior therapies, who were treated with DAC 0.15 mg/kg intravenously daily × 5 days/week for 2 weeks, TMZ orally 75 mg/m^2 qd for weeks 2-5 of a 6-week cycle.
Arm/Group | Dose Level 1:DAC (Decitabine) 0.075 mg/kg + TMZ (Temozolomide) | Dose Level 2:DAC (Decitabine) 0.15 mg/kg + TMZ (Temozolomide)
Number analyzed (Participants) | 2 | 6
percentage of participants | 0 | 17

2. Primary Outcome: Overall Response Rate (ORR)
Description: Using RECIST v1.0 criteria, overall response rate (ORR) was determined by the number of participants with complete response (CR) + the number of participants with partial response (PR) / the number of participants with complete response (CR) + the number of participants with partial response (PR) + the number of participants with stable disease (SD) + the number of participants with progressive disease (PD), multiplied by 100. Per RECIST v1.0 criteria (assessed by MRI or CT): Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response (PR) nor sufficient increase to to qualify for Progressive Disease (PD); PD, 20% increase in the sum if target lesion or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: Up to 30 months
Measure: Number; unit: percentage of participants
Groups:
- DAC (Decitabine) + TMZ (Temozolomide): Patients with non-resectable stage IIIB/C or stage IV metastatic melanoma with either no prior therapy or have progressed despite prior therapies, who were treated with Intravenous DAC of 0.15 mg/kg daily for 5 days a week for the first 2 weeks of a 6-week cycle who received TMZ orally at 75 mg/m^2 daily for 4 weeks (weeks 2-5) of a 6-week cycle.
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 33
percentage of participants | 18

3. Primary Outcome: Recommended Phase 2 Dose (RP2D) of DAC + TMZ
Description: Toxicity assessments used CTCAE v3.0. Two dose levels were explored in the phase I portion of the study. A modified 3 + 3 'up and down' design was used. Given the knowledge that DAC exhibits its epigenetic effects at 30-fold lower doses than at its maximum-tolerated dose (MTD), escalation of DAC to the MTD was not done.
Time Frame: Up to 26 months
Measure: Number; unit: mg/kg DAC
Arm/Group | Single Arm
Number analyzed (Participants) | 8
mg/kg DAC | 0.15

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Using RECIST v1.0 criteria, disease control rate (DCR) was determined by the number of participants with complete response (CR) + the number of participants with partial response (PR) + the number of participants with stable disease (SD) / the number of participants with complete response (CR) + the number of participants with partial response (PR) + the number of participants with stable disease (SD) + the number of participants with progressive disease (PD). Per RECIST v1.0 criteria (assessed by MRI or CT): Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response (PR) nor sufficient increase to to qualify for Progressive Disease (PD); PD, 20% increase in the sum if target lesion or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: Up to 30 months
Measure: Number; unit: percentage of participants
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 33
percentage of participants | 61

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from study entry until the documented radiological or symptomatic progression. Per RECIST v1.0 criteria (assessed by MRI or CT): Progressive Disease (PD); PD, 20% increase in the sum if target lesion or the appearance of new lesions.
Time Frame: Up to 42 months
Measure: Median (Full Range); unit: months
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 33
months | 3.4 [1.0 to 20.4]

6. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Time Frame: 6 months
Population: Patients that either progressed or died by 6 months.
Measure: Number; unit: percentage of participants
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 33
percentage of participants | 32.4

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from study entry until the death or date of last contract.
Time Frame: Up to 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 33
months | 12.4 [10.4 to 20.4]

8. Secondary Outcome: 1-year Overall Survival (OS) Rate
Description: Percentage of patients alive at one year (number of patients alive / total number of evaluable (analyzed) patients).
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Number analyzed (Participants) | 33
percentage of participants | 56

ADVERSE EVENTS:
Groups:
- DAC (Decitabine) + TMZ (Temozolomide): Comprehensive listing of adverse events are presented in total (includes events from both Phase 1 and and Phase 2 of study).
Arm/Group | DAC (Decitabine) + TMZ (Temozolomide)
Serious Adverse Events (participants affected / at risk) | 7/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DAC (Decitabine) + TMZ (Temozolomide) (N=39)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Febrile neutropenia (Infections and infestations) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Pain, Abdomen NOS (General disorders) | 2
Pain, Back (General disorders) | 1
Peripheral arterial ischemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAC (Decitabine) + TMZ (Temozolomide) (N=39)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 5
Anorexia (General disorders) | 15
Confusion (Nervous system disorders) | 3
Constipation (Gastrointestinal disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 10
Dizziness (Nervous system disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9
Edema: limb (Blood and lymphatic system disorders) | 10
Fatigue (asthenia, lethargy, malaise) (General disorders) | 35
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 5
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 8
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 3
Hypertension (Cardiac disorders) | 6
Infection with normal ANC or Grade 1 or 2 neutrophils, Skin (cellulitis) (Infections and infestations) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 3
Insomnia (General disorders) | 8
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 31
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 7
Mood alteration, Anxiety (Nervous system disorders) | 11
Mood alteration, Depression (Nervous system disorders) | 8
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 31
Neuropathy: sensory (Nervous system disorders) | 9
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 32
Pain, Abdomen NOS (General disorders) | 14
Pain, Back (General disorders) | 11
Pain, Chest wall (General disorders) | 3
Pain, Extremity-limb (General disorders) | 11
Pain, Head/headache (General disorders) | 17
Pain, Joint (General disorders) | 6
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Platelets (Blood and lymphatic system disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 8
Weight loss (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes